CLINICAL TRIAL: NCT03753308
Title: Mechanism of DCs Dysfunction in Chronic HBV Infection
Acronym: HepatoDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.198
Record Dates: First submitted 2018-11-23; First posted 2018-11-26 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: HBV; NASH - Nonalcoholic Steatohepatitis
Keywords: Dendritic cells; C-type lectins (CLR); mDCs BDCA1+ and BDCA3+ circulating and hepatic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1a, HBV patients / no scheduled biopsy: Intervention : Blood Sampling
  Eligibility criteria :
  * Male or female, Age of 18 or older, Weight over 40kg
  * Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
  * Patients who signed a non-opposition
  * Patient affiliated to social security insurance
  * HBsAg positive for more than 6 months
  * known status of HBeAg (positive or negative)
  * Treated or not with an antiviral
  Interventions: Biological: Blood Sampling
- 1b, HBV patients / with scheduled biopsy: Intervention : Liver biopsy
  Eligibility criteria :
  * Male or female, Age of 18 or older, Weight over 40kg
  * Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
  * Patients who signed a non-opposition
  * Patient affiliated to social security insurance
  * HBsAg positive for more than 6 months
  * known status of HBeAg (positive or negative)
  * Treated or not with an antiviral
  * Patient with a liver biopsy indication as part of the treatment within 3 months.
  Interventions: Biological: Liver biopsy
- 2, NASH patients / with scheduled biopsy: Intervention : Liver biopsy
  Eligibility criteria :
  * Male or female, Age of 18 or older, Weight over 40kg
  * Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
  * Patients who signed a non-opposition
  * Patient affiliated to social security insurance
  * The existence of at least one element of metabolic syndrome
  * Steatosis detected by non-invasive tests (echo, CAP, MRI)
  Interventions: Biological: Liver biopsy
- 3, Blood samples from healthy donors: * No subject will be included in this group, the samples have been already collected at EFS from healthy donors who had previously given their informed consents for using their blood samples in the research.
  * The blood samples have been collected in sufficient quantity to carry out the analyzes (20mL from each donor).
  Interventions: Biological: Blood Sampling

INTERVENTIONS:
Biological: Blood Sampling — 5 x Lithium Heparin Tubes WITHOUT DARK GREEN GEL, 5 ml- v. 4 ml Blood volumes collected as part of the usual care and this research comply with the recommendations of Jarde's law for an observational study (less than 80 ml in one day and less than 160 ml over 30 consecutive days for a subject over 40kg).
  Groups: 1a, HBV patients / no scheduled biopsy; 3, Blood samples from healthy donors
Biological: Liver biopsy — The liver biopsy is part of the usual care and it follows the usual procedure of CHUGA:
  The patient is placed in a supine position and received a transitory sedation, MEOPA gas (Kalinox®). Also, an ultrasound scan is performed. Local disinfection followed by local anesthesia with Xylocaine® are performed. The biopsy is performed with the Hepafix 17 gauge needle. 1 passage is carried out to obtain a biopsy fragment of at least 20 mm for the diagnosis (if the passage is unsuccessful, a second passage can be performed strictly as part of the usual care and not as part of research). If the biopsy is> 20 mm, a fragment of the excess biopsy specimen (10% or 2 mm) will be cut and used for research in groups 1b and 2. This division is performed by the clinician directly on the fresh specimen
  Groups: 1b, HBV patients / with scheduled biopsy; 2, NASH patients / with scheduled biopsy

SUMMARY:
This research is to better understand the functional impairments of Dendritic cells (DCs) in chronic HBV infection. Aim is to determine if the virus is able to bind to the C-type lectin receptor (CLRs) of DCs to modulate their functions, also, to define the role of viral components and the molecular mechanisms of DCs modulation by HBV. This project should provide a better understanding of the mechanisms by which the immune response is altered by HBV and the immunological control of the infection, and thus propose new immunotherapeutic strategies based on the restoration of DC functions by releasing of virally-induced inhibitions, compromising the infection chronicity

DETAILED DESCRIPTION:
Currently, chronic hepatitis B virus (HBV) infection therapies are limited to pegylated interferon alpha (Peg-IFNα) and nucleos(t)ide analogues (NUCs), alone or in combination. Even though they can reduce viremia level (circulating viral load), the loss of HBs antigen (HBsAg), which indicates functional clearance of the virus, is achieved in less than 10% of cases.

The absence of curative treatment to eliminate the infection justifies the need to define new targets and to develop new therapeutic strategies, with an immuno-therapeutic component.

Chronic HBV infection is associated with persistent and virally-induced immune deficiency. The immunological control of the infection seems essential to the functional clearance of the virus. The restoration of appropriate immune responses against the virus could prove to be a promising therapeutic strategy. However, the mechanisms in which HBV modulates immune function is still poorly understood.

Dendritic cells (DCs) have an essential role in immunity. They play a central role in the induction and regulation of immune responses. Also, they play a particularly crucial role in the induction and orientation of antiviral immunity due to their unique properties at the interface between innate and acquired immune responses. In several chronic viral infections, DCs appear defective. The immune responses induced in the early stages of infection seem to be a crucial guide on the progression of the infection into the resolution or the chronicity.

Objective of the investigators is to better understand the virus escape mechanism from immune control, particularly, to determine the mechanisms in which the virus modulates the functions of DCs, crucial for the subsequent orientation of antiviral immune responses, to define the molecular mechanisms of this inhibition and their consequences on the antiviral effectors functions, in order to propose new immunotherapeutic approaches that compromise the chronicity of the infection and treat the infection permanently and definitively.

Lastly, the investigators have shown that there are functional impairments in plasmacytoid DCs (pDCs) in patients with chronic hepatitis B, associated with a lack of cytotoxic activity of NK cells. The Subverting of pDCs in HBV patients could be related to IP-10 and HBsAg and HBeAg antigens or other viral components (infectious particles or circulating HBcAg). In addition, HBV was able to inhibit the production of IFNα by pDCs from healthy individuals in response to TLR9 agonists, by the presence of inhibitory CpG sequences in its genome. This mechanism would allow the virus to actively escape the innate immune response mounted by pDCs. Recently, investigators have found an alteration of lectin C-type receptor (CLR) expression on pDCs of HBV patients compared to healthy donors as well as a phenotypic and functional modulation in the 3 major subtypes of DCs (mDCs BDCA1 +, pDCs BDCA2 + and mDCs BDCA3 +) in the context of chronic HBV infection. These major subversions of DCs, crucial cells for subsequent orientation of antiviral immune responses, support the hypothesis that HBV might deflect immunity by impacting these cells.

In this clinical trial, investigators would like to pursue their research to better understand the functional impairments of DCs in chronic HBV infection, by defining if the virus is able to bind to the CLRs of DCs to modulate their functions, and by defining the role of viral components and the molecular mechanisms of DCs modulation by HBV. This project should provide a better understanding of the mechanisms of the immune response orientation by HBV and the immunological control of the infection, and thus propose new immunotherapeutic strategies based on the restoration of DC functions by releasing of virally-induced inhibitions, compromising the infection chronicity

ELIGIBILITY:
Inclusion Criteria :

Group 1a: HBV positive patients / no scheduled biopsy

* Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
* Patients who signed a non-opposition
* Patient affiliated to social security insurance
* HBsAg positive for more than 6 months
* known status of HBeAg (positive or negative)
* Treated or not with an antiviral

Group 1b: HBV positive patients / with scheduled biopsy

* Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
* Patients who signed a non-opposition
* Patient affiliated to social security insurance
* HBsAg positive for more than 6 months
* known status of HBeAg (positive or negative)
* Treated or not with an antiviral
* Patient with a liver biopsy indication as part of the treatment within 3 months.

Group 2: NASH patients / with scheduled biopsy

* Surveyed as part of their usual care in Hepato-Gastroenterology clinic at CHUGA
* Patients who signed a non-opposition
* Patient affiliated to social security insurance
* The existence of at least one element of metabolic syndrome
* Steatosis detected by non-invasive tests (echo, CAP, MRI)

Group 3: Blood samples from healthy donors

* No subject will be included in this group, the samples have been already collected at EFS from healthy donors who had previously given their informed consents for using their blood samples in the research.
* The blood samples have been collected in sufficient quantity to carry out the analyzes (20mL from each donor).

Exclusion Criteria:

For groups 1a, 1b and 2 (HBV or NASH patients):

* Positive serology for HCV, HDV, HTLV, HIV
* Active autoimmune diseases
* Immunosuppressive therapies
* Cancer <2 years
* Alcohol: male> 30g / day, female> 20g / day

Group 1a and 1b:

* NASH patients

Group 2:

* Positive HBsAg Group 3: Blood samples from healthy donors
* Positive serology for HCV, HTLV, HIV, HBV (in the sense of a positive HBsAg test).
* Risk of any infectious disease at the time of sample collection (including fever> 38 ° C over the past 15 days or recent contact with a person with a contagious disease).
* Autoimmune disease or immunosuppressive therapy at the time of sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 88 HBV patients (44 blood sampling, 44 liver biopsy), 44 NASH patients (liver biopsy)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-12-05 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Define the subversion mechanism of dendritic cells (DCs) by hepatitis B virus (HBV) | 4 years
  Differential expression of the tested molecules (DCIR, dectin 1, DEC205, DC-SIGN, Clec12a, CD206, CD207, Clec9a, CD32) on circulating and hepatic mDCs (BDCA1+ et BDCA3+) of HBV patients compared to controls (healthy donors for circulating DCs, or NASH patients for hepatic DCs)

SECONDARY OUTCOMES:
Demonstrate the correlations between immunological and clinical parameters | 4 years
  Identify of clinical evolution prognostic factors and determine significant correlations between measured immunological parameters and HBV infection parameters (plasma levels of HBV DNA, HBsAg, HBeAg, ALT)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LEROY, Pr, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No